CLINICAL TRIAL: NCT05484323
Title: Acute Effects of Cookies Containing 2.5 g Spirulina on Postprandial Glycemic and Insulin Responses: A Randomized Clinical Trial in Healthy Humans
Brief Title: Acute Effects of Cookies Containing 2.5 g Spirulina on Postprandial Glycemic and Insulin Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agricultural University of Athens (Other)
Responsible Party: Principal Investigator, Aimilia Papakonstantinou, Assistant Professor, Agricultural University of Athens
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: HRBD 50 12/10/2021
Record Dates: First submitted 2022-07-30; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Potential Abnormality of Glucose Tolerance; Appetitive Behavior; Blood Pressure
Keywords: blood glucose responses; spirulina; blood glucose concentrations; glycemic index
MeSH Terms: conditions — Appetitive Behavior | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: Crossover, double blind, randomized clinical trial
Who Masked: Participant, Investigator
Masking Description: double-blind both the participant and investigator were masked. A researcher not involved in data analyses was responsible for participant allocation and test food consumption
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Glucose as reference food (Experimental): Thirteen healthy participants (male: 4, female: 9) after 10-14h fast, consumed 50 g available carbohydrates from D-glucose, in different visits as reference food, tested two times; and 50 g available carbohydrates from white bread, tested two times; and 50 g available carbohydrates from cookies containing 0 and 2.5g spirulina, tested once, in different visits, along with 250 mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose and salivary insulin samples were taken at 0, 15, 30, 45, 60, 90 and 120 min postmeal. The first glucose and salivary insulin sample were taken exactly 15 min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: White bread; Diagnostic Test: Cookie containing 0 g spirulina; Other: Cookie containing 2.5 g spirulina
- White bread (Experimental): Thirteen healthy participants (male: 4, female: 9) after 10-14h fast, consumed 50 g available carbohydrates from D-glucose, in different visits as reference food, tested two times; and 50 g available carbohydrates from white bread, tested two times; and 50 g available carbohydrates from cookies containing 0 and 2.5g spirulina, tested once, in different visits, along with 250 mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose and salivary insulin samples were taken at 0, 15, 30, 45, 60, 90 and 120 min postmeal. The first glucose and salivary insulin sample were taken exactly 15 min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: White bread; Diagnostic Test: Cookie containing 0 g spirulina; Other: Cookie containing 2.5 g spirulina
- Cookie containing 0 g spirulina (Experimental): Thirteen healthy participants (male: 4, female: 9) after 10-14h fast, consumed 50 g available carbohydrates from D-glucose, in different visits as reference food, tested two times; and 50 g available carbohydrates from white bread, tested two times; and 50 g available carbohydrates from cookies containing 0 and 2.5g spirulina, tested once, in different visits, along with 250 mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose and salivary insulin samples were taken at 0, 15, 30, 45, 60, 90 and 120 min postmeal. The first glucose and salivary insulin sample were taken exactly 15 min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: White bread; Diagnostic Test: Cookie containing 0 g spirulina; Other: Cookie containing 2.5 g spirulina
- Cookie containing 2.5 g spirulina (Experimental): Thirteen healthy participants (male: 4, female: 9) after 10-14h fast, consumed 50 g available carbohydrates from D-glucose, in different visits as reference food, tested two times; and 50 g available carbohydrates from white bread, tested two times; and 50 g available carbohydrates from cookies containing 0 and 2.5g spirulina, tested once, in different visits, along with 250 mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose and salivary insulin samples were taken at 0, 15, 30, 45, 60, 90 and 120 min postmeal. The first glucose and salivary insulin sample were taken exactly 15 min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: White bread; Diagnostic Test: Cookie containing 0 g spirulina; Other: Cookie containing 2.5 g spirulina

INTERVENTIONS:
Other: Glucose as reference food — Thirteen healthy participants (male: 4, female: 9) after 10-14h fast, consumed 50 g available carbohydrates from D-glucose, in different visits as reference food, tested two times; and 50 g available carbohydrates from white bread, tested two times; and 50 g available carbohydrates from cookies containing 0 and 2.5g spirulina, tested once, in different visits, along with 250 mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose and salivary insulin samples were taken at 0, 15, 30, 45, 60, 90 and 120 min postmeal. The first glucose and salivary insulin sample were taken exactly 15 min after the first bite of food or drink.
Other: White bread — Thirteen healthy participants (male: 4, female: 9) after 10-14h fast, consumed 50 g available carbohydrates from D-glucose, in different visits as reference food, tested two times; and 50 g available carbohydrates from white bread, tested two times; and 50 g available carbohydrates from cookies containing 0 and 2.5g spirulina, tested once, in different visits, along with 250 mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose and salivary insulin samples were taken at 0, 15, 30, 45, 60, 90 and 120 min postmeal. The first glucose and salivary insulin sample were taken exactly 15 min after the first bite of food or drink.
Diagnostic Test: Cookie containing 0 g spirulina — Thirteen healthy participants (male: 4, female: 9) after 10-14h fast, consumed 50 g available carbohydrates from D-glucose, in different visits as reference food, tested two times; and 50 g available carbohydrates from white bread, tested two times; and 50 g available carbohydrates from cookies containing 0 and 2.5g spirulina, tested once, in different visits, along with 250 mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose and salivary insulin samples were taken at 0, 15, 30, 45, 60, 90 and 120 min postmeal. The first glucose and salivary insulin sample were taken exactly 15 min after the first bite of food or drink.
Other: Cookie containing 2.5 g spirulina — TThirteen healthy participants (male: 4, female: 9) after 10-14h fast, consumed 50 g available carbohydrates from D-glucose, in different visits as reference food, tested two times; and 50 g available carbohydrates from white bread, tested two times; and 50 g available carbohydrates from cookies containing 0 and 2.5g spirulina, tested once, in different visits, along with 250 mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose and salivary insulin samples were taken at 0, 15, 30, 45, 60, 90 and 120 min postmeal. The first glucose and salivary insulin sample were taken exactly 15 min after the first bite of food or drink.

SUMMARY:
This study investigated the effects of cookies containing 2.5 g Spirulina on postprandial glycemic and insulin responses.

DETAILED DESCRIPTION:
This study examined the short-term effects of cookies containing 0 and 2.5 g Spirulina on postprandial glycemic and insulin responses, arterial blood pressure and subjective appetite

ELIGIBILITY:
Inclusion Criteria:

* healthy
* non-smoking
* men and women
* body mass index between 18 and 24.9 kg/m2

Exclusion Criteria:

* severe chronic disease (e.g. cardiovascular diseases, diabetes mellitus, kidney or liver conditions, endrocrine conditions)
* gastrointestinal diseases
* pregnancy
* lactation
* competitive sports
* alcohol abuse
* drug dependency

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Capillary blood glucose responses | 2 hours
  Clinically useful change in blood glucose, defined as the restoration of glucose within normal limits during the 2 hr glucose tolerance test

SECONDARY OUTCOMES:
Salivary insulin responses | 2 hours
  Clinically useful change in salivary insulin, defined as the restoration of insulin within normal limits during the 2hr glucose tolerance test

OTHER OUTCOMES:
Subjective appetite ratings | 2 hours
  Useful change in subjective appetite using visual analogue scales with a score 0 to 10 (given in the form of booklet, one scale per page) at baseline, 15, 30, 45, 60, 90 and 120min. The minimum or maximum score will be evaluated if it is better or worse depending on the appetite variable e.g. hunger, satiety, desire to eat etc
Blood pressure | 2 hours
  Useful change in systolic and diastolic blood pressure before and 2hr after consumption of the cookie products

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Papakonstantinou, PhD, Principal Investigator — Agricultural University of Athens
Locations (1):
- Agricultural University of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: No